CLINICAL TRIAL: NCT03385759
Title: A Prospective Randomized Trial of Unicompartmental Versus Total Knee Arthroplasty for the Treatment of Medial Compartment Osteoarthritis
Brief Title: Trial of Unicompartmental Versus Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Anderson Orthopaedic Research Institute (Other)
Collaborators: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Nancy Parks, Sr. Project Director, Anderson Orthopaedic Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-2931
Record Dates: First submitted 2017-12-21; First posted 2017-12-28 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Osteo Arthritis Knee
Keywords: unicompartmental knee; total knee arthroplasty; osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- UKA (Active Comparator): Medial unicompartmental knee arthroplasty
  Interventions: Procedure: Unicompartmental knee arthroplasty
- TKA (Active Comparator): Total knee arthroplasty
  Interventions: Procedure: Total knee arthroplasty

INTERVENTIONS:
Procedure: Unicompartmental knee arthroplasty — Implant to replace the medial compartment of a patient with knee osteoarthritis
  Arms: UKA
Procedure: Total knee arthroplasty — Implant to replace the knee joint of a patient with knee osteoarthritis
  Arms: TKA

SUMMARY:
This study is a prospective, randomized trial to compare patient outcomes of unicompartmental knee arthroplasty (UKA) and total knee arthroplasty (TKA) for the treatment of medial compartment osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* medial compartment osteoarthritis of the knee
* knee flexion greater than greater than 90 degrees
* flexion contracture of less than 10 degrees
* varus deformity < 20 degrees
* grade IV degeneration of the medial compartment

Exclusion Criteria:

* lateral compartment degenerative changes
* previous lateral meniscectomy
* anterior cruciate ligament deficiency
* body mass index > 40
* inflammatory arthritis
* history of septic arthritis
* hemoglobin A1c > 8.0
* chronic liver disease
* stage 3A or greater chronic renal disease
* active IV drug abuse
* patients requiring thromboembolic prophylaxis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2018-05-22 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Knee Society Score | 1 year
  Functional outcome questionnaire ranging from 0-100, with 100 being best
Knee Society Score | 2 years
  Functional knee outcome questionnaire ranging from 0-100, with 100 being best

SECONDARY OUTCOMES:
Revision | 2 years
  complication requiring revision surgery

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Fricka, MD, Principal Investigator — Anderson Orthopaedic Institute
Locations (2):
- United States (2):
  - Rush University Medical Center, Chicago, Illinois
  - Anderson Orthopaedic Research Institute, Alexandria, Virginia

IPD SHARING:
Plan to Share IPD: No